CLINICAL TRIAL: NCT05650905
Title: Retinal Neurovascular Coupling in Patients Previously Infected With COVID-19
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Associate Professor, MD, PhD, Medical University of Vienna
Other Study IDs: OPHT-180520
Record Dates: First submitted 2022-12-13; First posted 2022-12-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; Post-COVID-19 Syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- subjects previously infected with COVID-19: subjects previously infected with COVID-19
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier domain optical coherence tomography (FDOCT); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG); Diagnostic Test: Proteomics and Metabolites in Plasma, tear fluid and finger sweat
- subjects with long COVID-19: subjects with long COVID-19 according to the WHO-guideline
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier domain optical coherence tomography (FDOCT); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG); Diagnostic Test: Proteomics and Metabolites in Plasma, tear fluid and finger sweat
- healthy age-and sex- matched control subjects with no history of COVID-19 infection: healthy age-and sex- matched control subjects with no history of COVID-19 infection
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier domain optical coherence tomography (FDOCT); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG); Diagnostic Test: Proteomics and Metabolites in Plasma, tear fluid and finger sweat

INTERVENTIONS:
Device: Dynamic Vessel Analyzer (DVA) — Retinal neurovascular coupling, Retinal vessel diameters and Retinal oxygen saturation will be assessed using the DVA
Device: Fourier domain optical coherence tomography (FDOCT) — Retinal blood velocities and Retinal blood flow will be assessed using the FDOCT
Device: Optical coherence tomography (OCT) — Retinal nerve fiber layer thickness, Central retinal thickness and Retinal vessel density will be assessed using the OCT
Device: Laser Speckle Flowgraphy (LSFG) — Normalized blur and Relative flow volume will be assessed using the LSFG
Diagnostic Test: Proteomics and Metabolites in Plasma, tear fluid and finger sweat — Proteomics and Metabolites in Plasma, tear fluid and finger sweat will be assessed using a Blooddraw, filter paper and Schirmer-test

SUMMARY:
The Study objective is to measure retinal neurovascular coupling and blood flow parameters in patients previously infected with COVID-19, long COVID-19 and healthy age- and sex- matched control subjects

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is affecting almost all countries in the world and because of its worldwide spread has been declared as pandemic in March 2020. While respiratory symptoms are the main manifestation of acute infection, there is also increasing evidence that neurological and vascular symptoms occur, and it is unknown whether residuals remain after patients have recovered. A recent report shows that changes in the human retina are even present one month after onset of symptoms. The eye, as an extension of the brain, offers the advantage that blood vessels as well as neural tissue can be visualized non-invasively in-vivo. Neurovascular coupling is the ability of neural tissue to adapt its blood flow to its metabolic demands, a phenomenon that does not only occur in the brain, but also in the retina. In the retina, neurovascular coupling can be studied by stimulating the retina with flicker light and measuring the response of the vessels. Retinal neurovascular coupling has been found to be impaired in diseases of the central nervous system (CNS) as well as in diseases associated with endothelial dysfunction. Since COVID-19 comes with CNS manifestations as well as endothelial dysfunction, we speculate that retinal neurovascular coupling might be impaired in patients even after they have recovered from COVID-19 infection. In the current study, retinal neurovascular coupling will be measured in patients who have recovered from COVID-19 infection with and without long COVID-19 and in healthy age- and sex-matched controls with no history of COVID-19 infection. In addition, retinal oxygen saturation, vessel diameters, vessel density as well as retinal and optic nerve head blood flow will be measured. To assess structural changes, measurement of central retinal thickness as well as retinal nerve fiber layer thickness will be performed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects

* Men and women aged over 18 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* No previous history of COVID-19 infection
* Negative testing for SARS-CoV-2 seroprevalence using nucleocapsid antibody tests
* Negative PCR test for SARS-CoV-2
* Normal ophthalmic findings, ametropy < 6 Dpt.

Inclusion criteria for subjects with history of COVID-19 infection

* Men and women aged over 18 years
* Non-smokers
* History of COVID-19 infection (confirmed by a positive PCR test for SARS-CoV2 in the medical history) within the last 6 months
* Positive testing for SARS-CoV-2 seroprevalence using spike protein IgG antibody tests
* Negative PCR test for SARS-CoV-2

Inclusion criteria for subjects with long COVID-19

* Men and women aged over 18 years
* Non-smokers
* History of COVID-19 infection (confirmed by a positive PCR test for SARS-CoV2 in the medical history)
* Positive testing for SARS-CoV-2 seroprevalence
* Negative PCR test for SARS-CoV-2
* Long Covid according to the latest WHO-Guidelines

Exclusion Criteria:

Any of the following will exclude a healthy control subject from the study:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Participation in a clinical trial in the 3 weeks preceding the study
* Blood donation during the previous three weeks
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Pregnancy, planned pregnancy or lactatin
* History of epilepsia

Any of the following will exclude a subject with history of COVID-19 infection from the study:

* Blood donation during the previous three weeks
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropy >6 Dpt
* Pregnancy, planned pregnancy or lactating
* History of epilepsia

Any of the following will exclude a subject with long COVID-19 from the study:

* Blood donation during the previous three weeks
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropy >6 Dpt
* Pregnancy, planned pregnancy or lactating
* History of epilepsia
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 90 subjects will be included:
  30 subjects previously infected with COVID-19 30 subjects with long COVID-19 30 age-and sex- matched subjects with no history of COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Retinal neurovascular coupling | Day 0
  Retinal neurovascular coupling will be assessed using the DVA

SECONDARY OUTCOMES:
Retinal vessel diameters | Day 0
  Retinal vessel diameters will be assessed using the DVA
Retinal oxygen saturation | Day 0
  Retinal oxygen saturation will be assessed using the DVA
Retinal blood velocities | Day 0
  Retinal blood velocities will be assessed using FDOCT
Retinal blood flow | Day 0
  Retinal blood flow will be assessed using FDOCT
Ocular perfusion pressure | Day 0
  Ocular perfusion pressure is going to be calulated
Retinal nerve fiber layer thickness | Day 0
  Retinal nerve fiber layer thickness will be assessed using OCT
Central retinal thickness | Day 0
  Central retinal thickness will be assessed using OCT
Retinal vessel density | Day 0
  Retinal vessel density will be assessed using OCT
Normalized blur | Day 0
  Normalized blur will be assessed using LSFG
Relative flow volume | Day 0
  Relative flow volume will be assessed using LSFG
Proteomics and Metabolites in Plasma | Day -14 to -1
  Proteomics and Metabolites in Plasma will be assessed through a Blood Sample
Proteomics and Metabolites in tear fluid | Day 0
  Proteomics and Metabolites in tear fluid will be assessed using Schirmer
Proteomics and Metabolites in finger sweat | Day 0
  Proteomics and Metabolites in finger sweat will be assessed using finger sweat filters

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pai V, Bileck A, Hommer N, Janku P, Lindner T, Kauer V, Rumpf B, Haslacher H, Hagn G, Meier-Menches SM, Schmetterer L, Schmidl D, Gerner C, Garhofer G. Impaired retinal oxygen metabolism and perfusion are accompanied by plasma protein and lipid alterations in recovered COVID-19 patients. Sci Rep. 2024 Apr 10;14(1):8395. doi: 10.1038/s41598-024-56834-4. PMID 38600099